CLINICAL TRIAL: NCT02221700
Title: A Pilot Study of Massage for Symptom Reduction in Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Massage Therapy in Reducing Chemotherapy-Induced Peripheral Neuropathy in Patients With Gastrointestinal or Breast Malignancies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: 2014-0250; NCI-2015-00386 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0250 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Malignant Breast Neoplasm; Malignant Digestive System Neoplasm; Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Peripheral Nervous System Diseases | interventions — Massage

ARMS (4):
- Group I (leg massage 3 x weekly for 4 weeks) (Experimental): Patients undergo massage therapy over 30 minutes to the affected legs at the foot and toes, ending at the knee, thrice weekly for 4 weeks.
  Interventions: Procedure: Massage Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (leg massage 2 x weekly for 6 weeks) (Experimental): Patients undergo massage therapy over 30 minutes to the affected legs at the foot and toes, ending at the knee, twice weekly for 6 weeks.
  Interventions: Procedure: Massage Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (head/neck/shoulder massage 3 x weekly for 4 weeks) (Experimental): Patients undergo massage therapy over 30 minutes to the head, neck, and shoulder thrice weekly for 4 weeks.
  Interventions: Procedure: Massage Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group IV (head/neck/shoulder massage 2 x weekly for 6 weeks) (Experimental): Patients undergo massage therapy over 30 minutes to the head, neck, and shoulder twice weekly for 6 weeks.
  Interventions: Procedure: Massage Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Massage Therapy — Undergo massage therapy
  Other Names: Massage
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies massage therapy in reducing chemotherapy-induced nerve problems (peripheral neuropathy) that may cause pain, numbness, tingling, swelling, or muscle weakness in different parts of the body in patients with gastrointestinal or breast malignancies. Massage therapy may help reduce chemotherapy-induced peripheral neuropathy symptoms and improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES; I. To compare completion rates of two massage treatment protocols (twice-weekly for 6 weeks versus three times weekly for 4 weeks) for patients with chronic, chemotherapy-induced peripheral neuropathy.

SECONDARY OBJECTIVES:

I. To determine the initial efficacy and effect size estimates of twice versus three times weekly site specific (lower extremity) massage versus alternate massage site (head/neck/shoulder) control groups at treating chronic, lower extremity chemotherapy-induced peripheral neuropathy.

II. To determine the initial efficacy and effect size estimates of massage on patient quality of life and functional performance tests.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP I: Patients undergo massage therapy over 30 minutes to the affected legs at the foot and toes, ending at the knee, thrice weekly for 4 weeks.

GROUP II: Patients undergo massage therapy over 30 minutes to the affected legs at the foot and toes, ending at the knee, twice weekly for 6 weeks.

GROUP III: Patients undergo massage therapy over 30 minutes to the head, neck, and shoulder thrice weekly for 4 weeks.

GROUP IV: Patients undergo massage therapy over 30 minutes to the head, neck, and shoulder twice weekly for 6 weeks.

After completion of study, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* All gastrointestinal malignancies where the patient received oxaliplatin for cancer treatment or breast malignancies where patients have received docetaxel or paclitaxel for cancer treatment
* Greater or equal to 6 months from last chemotherapy treatment
* Must understand and read English, sign a written informed consent, and follow protocol requirements
* Must be willing to come to MD Anderson Main Campus (Texas Medical Center) for intervention
* Lower extremity neuropathy per patient report attributable to oxaliplatin, docetaxel or paclitaxel (neurotoxic chemotherapeutic agent) as determined by patient history of neurotoxic agent administration and no history of other attributable causes such as diabetic neuropathy
* Patient self-report neuropathy score greater than or equal to 3 on a 0 to 10 numeric scale and/or grade 2 or 3 neuropathy (according to the National Cancer Institute Common Toxicity Criteria 4 point grading scale)
* Within 2 weeks prior to study enrollment the patient must be on a stable dose of medications for management of chemotherapy-induced peripheral neuropathy (CIPN) symptoms; for at least 2 weeks prior to enrollment stable dose is defined as:

  * No change in drug class
  * Increases or decreases that are less than or equal to 20% of the total dosage; all drug classes are allowed

Exclusion Criteria:

* Patients with previously diagnosed peripheral neuropathy pre-dating their neurotoxic chemotherapy administration or from causes other than chemotherapy
* Platelets less than 50,000 within 6 months prior to study enrollment or
* Neutrophil count less than 500 within 6 months prior to study enrollment
* Deep venous thrombosis (DVT) diagnosed within 12 months of study enrollment or history or untreated lower extremity DVT, bone metastases, currently active skin infection, or lymphedema currently involving the treatment field
* Women who are pregnant at time of enrollment; pregnancy will be assessed at enrollment using urine pregnancy test
* Diagnosis of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-04-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion Rates of Two Massage Treatment Protocols for Patients With Chronic, Oxaliplatin-Induced Peripheral Neuropathy | 10 weeks
  Completion rate defined as the average number of treatments completed of a possible 12 for patients in each protocol. Mean and standard deviation, along with a 95% confidence interval (CI) of the mean of the number of massages completed for each of the two massage schedules computed. Two-sample t-test used to compare the number of massages completed between the two schedules using a two-sided 0.05 significance level.

SECONDARY OUTCOMES:
Quality and intensity of neuropathic pain | At 10 weeks
  Will be measured by Pain Quality Assessment Scale (PQAS). To estimate the efficacy of the massage treatments at 10 weeks, linear regression will be used with PQAS as the dependent variable, massage site and schedule being two binary independent variables with interaction, adjusting for appropriate covariates such as the baseline value of PQAS. To assess the efficacy of the massage treatments over time linear mixed models (LMMs) will be used.
Quality of life (QOL) | Up to 10 weeks
  Will be measured by the Medical Outcomes Study Short Form 36. Pairwise comparisons between arms will be made as desirable, adjusting for multiple comparisons using the Bonferroni approach. Similar linear regression and LMM analyses will be carried out for the QOL and function measures.
Function and balance | Up to 10 weeks
  Will be measured by the Timed Up and Go test, the Single Limb Stance, and the Activities-Specific Balance Confidence Scale. Pairwise comparisons between arms will be made as desirable, adjusting for multiple comparisons using the Bonferroni approach. Similar linear regression and LMM analyses will be carried out for the QOL and function measures.
Symptoms associated specifically with chemotherapy-induced peripheral neuropathy | Up to 10 weeks
  Will be assessed using the Functional Assessment of Cancer Therapy/Gynecological Oncology Group-neurotoxicity version 4 questionnaire. Pairwise comparisons between arms will be made as desirable, adjusting for multiple comparisons using the Bonferroni approach. Similar linear regression and LMM analyses will be carried out for the QOL and function measures.
Baseline treatment expectations | Baseline
  Baseline treatment expectations will be assessed as a predictor of the secondary measures at week 10.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Lopez, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org